CLINICAL TRIAL: NCT05871983
Title: Clinical Evaluation of Safety and Effectiveness of the Munich Transcatheter Mitral Valve Replacement (TMVR) System
Brief Title: Munich Transcatheter Mitral Valve Safety and Effectiveness
Acronym: MUSE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: P+F Products + Features GmbH (Industry)
Collaborators: Meditrial USA Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP-MIT-001
Record Dates: First submitted 2023-04-11; First posted 2023-05-23 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Mitral Regurgitation; Mitral Valve Disease
Keywords: mitral regurgitation; heart failure
MeSH Terms: conditions — Mitral Valve Insufficiency; Heart Failure

STUDY DESIGN:
Intervention Model Description: This is a prospective, non-randomized, single-arm, international, multicenter, clinical study designed to evaluate the safety and performance of the P&F MUNICH TMVR System in a population of patients with moderate to severe symptomatic mitral regurgitation, who are not suitable for surgical or approved percutaneous treatments. All patients will be followed closely up to 12 months after the intervention and long-term safety and effectiveness will be collected annually up to 5 years.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-Arm (Experimental): This is a prospective, non-randomized, single-arm, international, multicenter, clinical study designed to evaluate the safety, efficacy, and performance of the P&F MUNICH TMVR System in a population of patients with moderate to severe symptomatic Mitral Regurgitation.
  Interventions: Device: MUNICH TRANSCATHETER MITRAL VALVE REPLACEMENT SYSTEM

INTERVENTIONS:
Device: MUNICH TRANSCATHETER MITRAL VALVE REPLACEMENT SYSTEM — The replacement valve consists of a self-expanding, tri-leaflet, dry bovine -pericardial valve. The dry tissue allows the valve to be conveniently pre-loaded. The key characteristics of Munich valve are:
  * Nitinol stent frame
  * Bovine pericardium
  * Polyester skirt
  * Anchoring system allows anchoring the frame to the annulus
  * Hooks are used to reduce the mobility of the native leaflets and decrease risk of embolization.
  The Munich TMVR system design proposed for this clinical investigation represents a significant evolution from previous TMVR designs:
  * Transfemoral / transseptal access
  * Self-expanding
  * Dry pericardium (can be pre-loaded)
  * No anchors
  * 27 Fr delivery catheter (
  * Sizes: 40/48/55mm
  * Height 30 mm The valve is available in 3 sizes with a 30mm profile and has been designed to reduce the complexity of implantation in comparison to other TMVR systems.

SUMMARY:
The Munich Trascatheter Mitral Valve System is intended for beating heart, mitral valve replacement in patients with a diseased, damaged, or malfunctioning mitral valve. Access is provided through the Femoral Vein and transseptal approach by means of a 27Fr catheter.

The bioprosthetic valve consists of a self-expanding, tri-leaflet, dry bovine-pericardial valve. The dry tissue allows the valve to be conveniently pre-loaded. The valve is available in three sizes and has been designed to reduce the complexity of implantation in comparison to other TMVR systems.

DETAILED DESCRIPTION:
This is a prospective multicenter clinical investigation designed to evaluate the safety and effectiveness of the Munich TMVR System in a population of patients with moderate to severe, symptomatic mitral regurgitation, who are not suitable for surgical treatments.

Patients who meet all of the study inclusion criteria, will be treated with the Munich valve. After the intervention, patients will be followed up closely for 12 months. Long term safety and efficacy data will be collected annually up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Moderate or severe mitral regurgitation (> 3+)

   1. For Degenerative MR: EROA ≥ 40 mm2 or regurgitant volume ≥ 60ml
   2. For Secondary MR: EROA > 30 mm2 or regurgitant volume > 45ml (i.e., MR moderate or severe by ASE criteria)
3. New York Heart Association (NYHA) Functional Class II, III or ambulatory IV
4. Subject is under guideline directed medical therapy for at least one month
5. Subject is high-risk for open-heart surgery based on the assessment of the multidisciplinary Heart Team using standard scoring systems and consideration of co-morbidities, frailty and disability
6. Subject meets the anatomical criteria for Munich TMVR System
7. Patient is willing to participate in the study and provides signed informed consent.

Exclusion Criteria:

General Conditions

1. Subject who is currently participating in an investigational study, other than this study
2. Subjects allergic to bovine tissue
3. Subjects with uncontrolled hypotension
4. Hemodynamic instability
5. Subject has contrast agent hypersensitivity that cannot be adequately pre-medicated and has an allergy to Nitinol alloys
6. Intolerance to antiplatelet, anticoagulant or thrombolytic medications
7. Bleeding diathesis or hypercoagulable state
8. Active peptic ulcer or active gastrointestinal bleeding
9. Pulmonary artery systolic pressure >70 mmHg
10. Renal insufficiency
11. Need for emergent or urgent surgery for any reason or any planned cardiac surgery within the next 12 months.
12. Subject with hepatic insufficiency
13. Subject has a co-morbid illness that may result in a life expectancy of less than one year
14. Active infection that requires antibiotic therapy
15. Subject is pregnant, breastfeeding or intend to become pregnant within one year, and female subjects in childbearing age NOT using a highly effective method of contraception with a failure rate of less than 1% per year.

    Comorbidities
16. Prior stroke or TIA within 3 months or Modified Rankin Scale ≥4 disability
17. Acute myocardial infarction within the previous 30 day
18. Any prior heart valve surgery or transcatheter mitral intervention
19. Any percutaneous cardiovascular intervention, cardiovascular surgery, or carotid surgery within 30 days
20. Rheumatic heart disease or endocarditis within the previous 3 months
21. Hypertrophic cardiomyopathy, restrictive cardiomyopathy, constrictive pericarditis
22. Severe organic lesion with retracted chordae or congenital malformation and lack of valvular tissue
23. Any other structural heart disease causing heart failure other than dilated cardiomyopathy of either ischemic or non-ischemic etiology.
24. Existence of inferior vena cava filter or atrial septal device (contraindicating femoral access and transseptal catheterization)
25. Untreated clinically significant coronary artery disease requiring revascularization
26. Tricuspid valve disease requiring surgery or severe tricuspid regurgitation
27. Aortic or pulmonic valve disease requiring surgery
28. CRT/ICD implant within 30 days
29. NYHA class IVb
30. UNOS stadium 1 heart transplantation or previous orthotopic heart transplantation

    Anatomical and Functional
31. Left Ventricular Ejection Fraction (LVEF) <30%
32. LV end diastolic diameter > 70mm
33. Significant abnormalities of the sub-valvular apparatus.
34. Severe mitral annular or leaflets calcification
35. Left atrial or LV thrombus or vegetation
36. Severe right ventricular dysfunction
37. Severe tricuspid or aortic valve disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07-30 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoints | 30 days
  The primary safety endpoint is to evaluate a 30-day major adverse events (MAE) rate, where MAE is a composite of the following device- or procedure-related events:
  * All-cause mortality
  * Stroke
  * Life-threatening bleeding (MVARC scale)
  * Major vascular complications
  * Major cardiac structural complications
  * Myocardial infarction or coronary ischemia requiring PCI or CABG
  * Stage 2 or 3 acute kidney injury (includes new dialysis)
  * Severe hypotension, worsening of heart failure, or respiratory failure requiring intravenous pressor or invasive or mechanical heart failure treatments such as ultraﬁltration or hemodynamic assist devices, including intra-aortic balloon pumps or left ventricular or biventricular assist devices, or prolonged intubation for >48 h.
  * Emergency surgery or re-intervention.

SECONDARY OUTCOMES:
Secondary Safety Endpoints | 90-day, 180-day, 1 year and annually at year 2, 3, 4 and 5
  Secondary safety endpoints include an evaluation at 90-day, 180-day, 1 year and annually at year 2, 3, 4 and 5 (inclusive of unscheduled visits):
  * Death, cardiac, non-cardiac
  * Stroke
  * Myocardial Infarction
  * Any device related complication/ dysfunction
  * New atrial fibrillation (AF)
  * New conduction disturbance requiring permanent pacemaker (PM)
  * Major access and vascular complications
  * Stage 2 or 3 acute kidney injury (includes dialysis)
  * Any valve-related dysfunction, migration, thrombosis, or other complication requiring surgery or repeat intervention

OTHER OUTCOMES:
Secondary Performance Assessment | Intraprocedural
  Technical success of the procedure, defined as successful access to the left atrium, delivery and deployment of the Munich Valve in the correct position and retrieval of delivery catheter, without significant mitral stenosis, LVOT obstruction or paravalvular MR documented by intraoperative imaging.
Secondary Effectiveness Assessment: Reduction of mitral regurgitation | 30-day, 90-day, 180-day, 1-year and annually at year 2, 3, 4,5
  Reduction of mitral regurgitation (MR) to either optimal (0+ to trace) or acceptable
Secondary Effectiveness Assessment: Changes in Ejection Fraction | 30-day, 90-day, 180-day, 1-year and annually at year 2, 3, 4,5
  Changes in Ejection Fraction
Secondary Effectiveness Assessment: NYHAC | 30-day, 90-day, 180-day, 1-year and annually at year 2, 3, 4,5
  New York Heart Association Class
Secondary Effectiveness Assessment: KCCQ | 30-day, 90-day, 180-day, 1-year and annually at year 2, 3, 4,5
  Quality of Life Improvement vs. Baseline (Kansas City Cardiomyopathy Questionnaire, KCCQ - Appendix I)
Secondary Effectiveness Assessment: Hospitalization Rate | 30-day, 90-day, 180-day, 1-year and annually at year 2, 3, 4,5
  Rate of hospitalizations for heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Katharina Kiss, MD, Study Chair — CEO, Products & Features
Locations (10):
- Argentina (4):
  - Fundación Favaloro, Buenos Aires
  - Hospital Italiano De Buenos Aires, Buenos Aires
  - Hospital César Milstein, Buenos Aires
  - Hospital Fernandez/Sanatorio Milstein, Buenos Aires
- Brazil (3):
  - Instituto Estadual De Cardiologia Aloysio De Castro, Rio de Janeiro
  - Instituto Dante Pazzanese De Cardiologia, São Paulo
  - Instituto Do Coração (InCor) De São Paulo, São Paulo
- Chile (3):
  - Hospital Del Torax De Santiago, Santiago
  - Hospital Dr Sotero Del Rio De Santiago, Santiago
  - Hospital Las Higueras - Talcahuano, Talcahuano

REFERENCES:
- See also: Products & Features, manufacturer of MUNICH Transcatheter Mitral Valve System — https://productsandfeatures.com/
- See also: Meditrial Clinical Research Organization — http://meditrial.net